CLINICAL TRIAL: NCT03027284
Title: A Phase I Study of Merestinib Monotherapy or in Combination With Other Anti-Cancer Agents in Japanese Patients With Advanced and/or Metastatic Cancer
Brief Title: A Study of Merestinib (LY2801653) in Japanese Participants With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16330; I3O-JE-JSBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05-15

CONDITIONS: Advanced Cancer; Metastatic Cancer; Biliary Tract Carcinoma; Cholangiocarcinoma; Gall Bladder Carcinoma; Solid Tumor; Non-Hodgkin's Lymphoma
Keywords: Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Cholangiocarcinoma; Gallbladder Neoplasms; Lymphoma, Non-Hodgkin; Neoplasms | interventions — merestinib; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Merestinib (Part A Dose Level 1) (Experimental): Merestinib administered orally. Treatment will continue until disease progression, development of unacceptable toxicity, or other discontinuation criteria are met.
  Interventions: Drug: Merestinib
- Merestinib (Part A Dose Level 2) (Experimental): Merestinib administered orally. Treatment will continue until disease progression, development of unacceptable toxicity, or other discontinuation criteria are met.
  Interventions: Drug: Merestinib
- Merestinib + Cisplatin + Gemcitabine (Part B) (Experimental): Merestinib administered orally with cisplatin and gemcitabine administered intravenously (IV). Treatment will continue until disease progression, development of unacceptable toxicity, or other discontinuation criteria are met, but Cisplatin and gemcitabine treatment will be limited to a maximum of 8 cycles.
  Interventions: Drug: Merestinib; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Merestinib — Administered orally
  Other Names: LY2801653
Drug: Cisplatin — Administered IV
  Arms: Merestinib + Cisplatin + Gemcitabine (Part B)
Drug: Gemcitabine — Administered IV
  Other Names: LY188011
  Arms: Merestinib + Cisplatin + Gemcitabine (Part B)

SUMMARY:
The main purpose of this study is to evaluate tolerability of merestinib monotherapy or in combination with other anti-cancer agents in Japanese participants with advanced and/or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic (solid tumors or non-Hodgkin's lymphoma).
* Part B: Biliary tract carcinoma that is unresectable, recurrent, or metastatic. The participant must not have received prior systemic front-line therapy for metastatic or resectable disease.
* Part A: Measurable or nonmeasurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Cheson Criteria.
* Part B: Measurable disease as defined by RECIST v1.1.
* Adequate organ function including hematologic, hepatic and renal.
* Eastern Cooperative Oncology Group (ECOG) scale of 0 or 1.
* Are able to swallow tablets.
* For participants in Part B, a tumor tissue sample is mandatory for biomarker analysis.
* Males must agree to use medically approved barrier contraceptive precautions during the study and for 3 months following the last dose of study drug.
* Females with childbearing potential: Must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug, must have had a negative serum or urine pregnancy test ≤7 days before the first dose of study drug.
* A breastfeeding woman must not be breastfeeding. If a female who stops breastfeeding enters the study, breastfeeding must cease from the day of the first study drug administration until at least 3 months after the last administration.

Exclusion Criteria:

* Have serious pre-existing medical conditions.
* Have a chronic underlying infection.
* Have symptomatic central nervous system malignancy or metastasis.
* Have an active fungal, bacterial, and/or known viral infection.
* Part B: Have mixed hepatocellular biliary tract carcinoma histology.
* Have liver cirrhosis with a Child-Pugh stage of B or higher, or have received a liver transplant.
* Have a history of congestive heart failure with New York Heart Association (NYHA) class greater than 2, unstable angina, or have recent history of myocardial infarction, transient ischemic attacks, stroke, or arterial or venous vascular disease.
* Have a corrected QT interval >470 milliseconds as calculated be the Fredericia equation.
* Have a second primary malignancy that, in the judgment of the investigator, and sponsor may affect the interpretation of results.
* Have any evidence of clinically active interstitial lung disease (ILD).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Merestinib Dose-Limiting Toxicities (DLTs) | Cycle 1 (Part A = 28 Days or Part B = 21 Days)
  Number of participants with DLTs

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Merestinib and its Metabolites | Predose Cycle 1 Throughout the First 2 Cycles (Part A = 28-Day Cycles, Part B = 21-Day Cycles)
  PK: Cmax of merestinib and its metabolites
PK: Area Under the Concentration Time Curve (AUC) of Merestinib and its Metabolites | Predose Cycle 1 Throughout the First 2 Cycles (Part A = 28-Day Cycles, Part B = 21-Day Cycles)
  PK: AUC of merestinib and its metabolites
Objective Response Rate (ORR): Percentage of Participants With a Complete or Partial Response | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Estimated as up to 8 Months)
  ORR: Percentage of participants with a complete or partial response
Disease Control Rate (DCR): Percentage of Participants with a Best Overall Response of Complete Response, Partial Response, and Stable Disease | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Estimated as up to 8 Months)
  DCR: Percentage of participants with a best overall response of complete response, partial response, and stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tokyo

REFERENCES:
- [Derived] Doi T, Yamamoto N, Naito Y, Kuboki Y, Koyama T, Piao Y, Tsujimoto N, Asou H, Inoue K, Kondo S. Merestinib monotherapy or in combination for japanese patients with advanced and/or metastatic cancer: A phase 1 study. Cancer Med. 2021 Oct;10(19):6579-6589. doi: 10.1002/cam4.4110. Epub 2021 Sep 9. PMID 34499416